CLINICAL TRIAL: NCT02820077
Title: Randomized Controlled Trial of Hemostatic Powder Versus Optimal Clinical Management for the Treatment of Upper Gastrointestinal Bleeding From Tumor Lesions
Brief Title: Hemostatic Powder Versus Clinical Management for the Treatment of Upper Gastrointestinal Bleeding From Tumor Lesions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Global recall of Hemospray
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Fauze Maluf Filho, Professor, Instituto do Cancer do Estado de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP883/15
Record Dates: First submitted 2016-06-07; First posted 2016-06-30 (Estimated); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Gastrointestinal Hemorrhage; Gastrointestinal Neoplasms
Keywords: Endoscopy, Gastrointestinal
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Gastrointestinal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemospray (Experimental): Patients treated with hemostatic powder
  Interventions: Device: Hemospray (Endoscopic treatment with hemostatic powder)
- Clinical support (No Intervention): Patients treated with optimal clinical management, as it is been advised by the latest guidelines

INTERVENTIONS:
Device: Hemospray (Endoscopic treatment with hemostatic powder) — Malignant bleeding lesions will be treated with endoscopic powder and patients will receive optical clinical management afterwards
  Arms: Hemospray

SUMMARY:
This study evaluates the efficacy of the endoscopic hemostatic powder for the treatment of bleeding from malignant lesions of the upper GI tract. Half of participants will receive hemostatic powder and half will be submitted to standard treatment.

DETAILED DESCRIPTION:
Gastrointestinal tumor bleeding is a challenging clinical condition with a high mortality rate. Several endoscopic hemostasis techniques have been tested, but results were disappointing. Re-bleeding and mortality rates are still high.

Hemostatic powder is a promising therapy for tumor bleeding, since it can be applied over large surfaces. Bleeding from a tumor lesion often occurs diffusely on the surface of the tumor rather than from a specific vessel.

ELIGIBILITY:
Inclusion Criteria:

* Any kind of malignancy
* Gastrointestinal bleeding in the last 48 hours
* Referred to emergency endoscopy

Exclusion Criteria:

* under 18 years old
* bleeding from non malignant lesions
* previous endoscopic treatment with another method done in the last 48h

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-08-06 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
rebleeding | until 30 days after endoscopy
mortality | until 30 days after endoscopy

SECONDARY OUTCOMES:
Successful initial hemostasis | From the moment of the procedure until 24 hours after it
Hospital length of stay | from the moment of the endoscopic procedure until hospital discharge or death, whichever came first, assessed up to 100 months

IPD SHARING:
Plan to Share IPD: No